CLINICAL TRIAL: NCT03909828
Title: Precision Medical Diagnosis and Acupuncture Treatment for Parkinson's Disease - The Quantitative Analysis System for PET/MRI Images in Patients
Brief Title: Precision Medical Diagnosis for Parkinson's Disease - The Quantitative Analysis System for PET/MRI Images in Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-10-001B
Record Dates: First submitted 2019-01-22; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Parkinson Disease; PET; MRI
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's disease patients: patients with Idiopathic Parkinsonism

SUMMARY:
In nuclear medicine PET examinations, labeled radiopharmaceuticals are possible to enter the putamen and caudate nucleus regions of the striatum in the brain by intravenous injection. The severity of Parkinson's disease is assessed and diagnosed by quantitative analysis of the defect in the image of the radiopharmaceuticals. Clinical studies often use manual selection of regions of interest (ROIs) for quantitative analysis. However, this method causes human error and low reproducibility due to subjective factors, and also considerable time consuming. Therefore, in order to solve the above problems, this research project plans to build an automated quantitative analysis system for PET/MRI images. The quantitative analysis of the PET images is performed automatically by using the putamen and caudate ROI segmented by the MRI images. This automated quantitative analysis system is expected to improve the time-consuming, low reproducibility, and subjectivity problems of traditional manual ROI selection method, and provide a useful tool for the diagnosis of early PD. In the first year, this sub-project is expected to perform MRI T1 and 18F-FDOPA PET scanning of before and after acupuncture-treated PD patients provided by sub-project 3. In the second year, the correlation analysis will be made with the results of tremor test provided by sub-project 1 and that of the 99mTc-TRODAT SPECT image quantification provided by sub-project 4.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disease whose pathogenic mechanism is the degeneration of substantia nigra of the midbrain, causing the degeneration of dopaminergic neurons in the putamen and caudate nucleus of the striatum, and the dopamine content in the synapses decreases and gradually loses the ability to act. Most of the clinical symptoms are motor function defects. The most obvious symptoms are tremor, limb stiffness, motor dysfunction and gait abnormality, and cognitive and behavioral problems may occur. In nuclear medicine PET examinations, labeled radiopharmaceuticals are possible to enter the putamen and caudate nucleus regions of the striatum in the brain by intravenous injection. The severity of Parkinson's disease is assessed and diagnosed by quantitative analysis of the defect in the image of the radiopharmaceuticals. Clinical studies often use manual selection of regions of interest (ROIs) for quantitative analysis. However, this method causes human error and low reproducibility due to subjective factors, and also considerable time consuming. Therefore, in order to solve the above problems, this research project plans to build an automated quantitative analysis system for PET/MRI images. The quantitative analysis of the PET images is performed automatically by using the putamen and caudate ROI segmented by the MRI images. In this study, patients will perform MRI T1 and 18F-FDOPA PET scanning of before and after acupuncture-treated PD patients in VGHTPE PET/MRI scanner. Every patient will be administered 185 MBq (5 mCi) of 18F-FDOPA by IV injection. The MRI image is used to extract the target and background ROIs (region of interests), and is coregistered to the PET image. The ROIs generated by MRI image will be applied to its corresponding PET image. Then, specific uptake ratio (SUR) will be calculated for each patient. The calculation of SUR is the difference between the average image pixel value of the target ROI (left and right striatum) and the average image pixel value of the background ROI (occipital lobe) divided by the average value of the background ROI. After calculated each patients' standard uptake ration, Asymmetry index (ASI) can be calculated based on the absolute difference of SUR value of both sides (left and right) of striatum, divided by average SUR value of both sides of striatum. This automated quantitative analysis system is expected to improve the time-consuming, low reproducibility, and subjectivity problems of traditional manual ROI selection method, and provide a useful tool for the diagnosis of early PD. In the first year, this sub-project is expected to perform MRI T1 and 18F-FDOPA PET scanning of before and after acupuncture-treated PD patients provided by sub-project 3. In the second year, the correlation analysis will be made with the results of tremor test provided by sub-project 1 and that of the 99mTc-TRODAT SPECT image quantification provided by sub-project 4.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as Idiopathic Parkinsonism by Neurologist
2. Have taken first line drugs more than three months
3. Did not take any acupuncture or rehabilitation
4. Voluntary

Exclusion Criteria:

1. Taking anticancer drug now or diagnosed as depression, psychosis or other mental illnesses
2. Medical history of stroke or dementia
3. Taking anticoagulant now or having coagulation disorders
4. Scalp infection
5. Pregnant women
6. Patient with irregular heartbeat, implanted artificial cardiac pacemaker or implanted cardioverter-defibrillator
7. Belonephobia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population consist of the participants who fulfill the inclusion criteria in eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The comparison of the change of Standard Uptake Ration (SUR) | 2 Months
  This study will collect images from a total of 100 PD patients (20 patients in the first year and 80 patients in the second year). Patients will perform MRI T1 and 18F-FDOPA PET scanning of before and after acupuncture-treated PD patients in VGHTPE PET/MRI scanner. Every patient will be administered 185 MBq (5 mCi) of 18F-FDOPA by IV injection. The MRI image is used to extract the target and background ROIs (region of interests), and is coregistered to the PET image. The ROIs generated by MRI image will be applied to its corresponding PET image. Then, specific uptake ratio (SUR) will be calculated for each patient. The calculation of SUR is the difference between the average image pixel value of the target ROI (left and right striatum) and the average image pixel value of the background ROI (occipital lobe) divided by the average value of the background ROI.The unit of pixel is mm and the unit of SUR measurement is percentage (%).

SECONDARY OUTCOMES:
The comparison of the change of asymmetry index (ASI) | 2 Months
  After calculated each patients' standard uptake ration, Asymmetry index (ASI) can be calculated based on the absolute difference of SUR value of both sides (left and right) of striatum, divided by average SUR value of both sides of striatum. The unit of ASI measurement is percentage (%).
Unified Parkinson's Disease Rating Scale | 2 Months
  A comprehensive assessment of both motor and non-motor symptoms associated with Parkinson's. The Unified Parkinson's Disease Rating Scale is made up of 42 items. These items are divided into six sections which are separately "evaluation of mentation, behavior, and mood", "self-evaluation of the activities of daily life", "clinician-scored monitored motor evaluation", "complications of therapy", "Hoehn and Yahr staging of severity of Parkinson's disease" and "Schwab and England ADL scale".The evaluation score for the first item to the 39th item is 0 to 4 points. The evaluation score for the 40th to the 42th item is 0 to 1 points. The higher score meand the worse condition. The sum of all the items'score is the score of the scale. Highr Rating Scales'scores indicate severe symptoms.
Micro Vibration Scan | 2 Months
  1. Discover early symptom before the onset.
  2. Recognize PD tremor pattern within 1 minute.
  3. Non-invasive, Non-radiation, and Low-cost medical device for daily tracking and treatment evaluation.
  1. Discover early symptom before the onset. 2. Recognize PD tremor pattern within 1 minute. 3. Non-invasive, Non-radiation, and Low-cost medical device for daily tracking and treatment evaluation.
  1. Discover early symptom before the onset.
  2. Recognize PD tremor pattern within 1 minute.
  3. Non-invasive, Non-radiation, and Low-cost medical device for daily tracking and treatment evaluation.
Constitution in Chinese Medicine Questionnaire (CCMQ) | 2 Months
  Sixty items were applied to measure the nine constitutions: Neutral (a normal constitution), Qi-deficiency constitution, Yang-deficiency constitution, Yin-deficiency constitution, Phlegm-dampness constitution, Damp-heat constitution, Stagnant-blood constitution, Stagnant-Qi constitution, and Inherited-special constitution.
Sphygmograph | 2 Months
  Diagnoses patient's pulse change

OTHER OUTCOMES:
statistical method-T test | 1 year
  after all the measure, we will use T test as the statistical method to do data analysis